CLINICAL TRIAL: NCT03821012
Title: China STEMI Care Project: a 10-year Project to Improve Quality of Care by Building up the a Regional STEMI Care Network
Brief Title: China STEMI Care Project
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yong Huo, Director, Department of Cardiology, Peking University First Hospital
Other Study IDs: CSCAP
Record Dates: First submitted 2019-01-22; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: ST-Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CSCAP-1: STEMI with symptom onset within 12 h regardless of whether receiving reperfusion or symptom onset within 12-24 h of needing PPCI
  Interventions: Other: in-hospital process optimization
- CSCAP-2: STEMI patients with symptom onset within 30 days
  Interventions: Other: PPCI hospital-based regional STEMI transfer network construction
- CSCAP-3: STEMI patients with symptom onset within 30 days
  Interventions: Other: the whole-city STEMI care network construction

INTERVENTIONS:
Other: in-hospital process optimization
  Groups: CSCAP-1
Other: PPCI hospital-based regional STEMI transfer network construction
  Groups: CSCAP-2
Other: the whole-city STEMI care network construction
  Groups: CSCAP-3

SUMMARY:
The China ST-elevation myocardial infarction (STEMI) Care Project (CSCAP) aims to improve the reperfusion treatment rate and shorten the total duration of myocardial ischemia by establishing a regional STEMI treatment network covering the whole-city region, whole-city population, and whole-disease process step by step. The CSCAP is a prospective, multicenter registry involving three phases. A total of 18 provinces, 4 municipalities, and 2 autonomous regions in China were included. Patients with STEMI who met with the third acute myocardial infarction definition and the Chinese STEMI diagnosis and treatment guidelines were enrolled and the estimated number is over 50,000. Phase 1 (CSCAP-1) focused on the in-hospital process optimization of primary percutaneous coronary intervention (PPCI) hospitals. Phase 2 (CSCAP-2) focused on the PPCI hospital-based regional STEMI transfer network, including emergency medical services and non-PPCI hospitals. Phase 3 (CSCAP-3) focused on the whole-city STEMI care network construction by promoting chest pain center accreditation. Systematic data collection, assessment of quality of care, and subsequent improvement were implemented throughout the project to continuously improve the quality of care for patients with STEMI.

CSCAP is the first project that focused on establishing a regional STEMI emergency care network in China to help understand the condition of STEMI care in China extensively. Moreover, its objective was to optimize the quality of STEMI care through in-hospital process optimization (2012-2013), PPCI hospital-based regional STEMI transfer network construction (2015-2018), and construction of the whole-city STEMI care network step by step (2018-2021). However, hospitals were not randomly selected in CSCAP, which might be because of the lack of representatives to some degree. Alternatively, it focused on providing a tailored quality-of-care improvement plan based on the conditions of different regions.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In CSCAP-1, a total of 4191 patients admitted to hospitals, with symptom onset within 12 h, regardless of whether receiving reperfusion or symptom onset within 12-24 h of needing PPCI, were enrolled consecutively in 53 tertiary hospitals qualified for PPCI in 14 provinces/municipalities/autonomous regions of China in 2012.
  In CSCAP-2, a total of 20,799 patients with STEMI occurrence within 30 days, regardless of reperfusion, were enrolled consecutively from PPCI hospitals 3 times at a 6-month interval in 244 PCI hospitals with hundreds of adjunct non-PCI hospitals from 24 provinces/municipalities/autonomous regions from 2015 to 2018.
  In CSCAP-3, a total of 30 hospitalized patients with symptom onset within 30 days were enrolled consecutively from each hospital every 3 months. Patients with STEMI were enrolled consecutively from the whole network units, including both PCI and non-PCI hospitals in 7 cities in China.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
the total duration of myocardial ischemia | 12 hours
  Median time from symptom onset to target vessel open in STEMI patients
the reperfusion treatment ratio | 12 hours
  the ratio of primary PCI plus thrombolysis usage in STEMI patients

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang Y, Yu B, Han Y, Wang J, Yang L, Wan Z, Zhang Z, Chen Y, Fu X, Gao C, Li B, Chen J, Wu M, Ma Y, Zhao X, Chen Y, Yan H, Xiang D, Fang W, Mehta S, Naber CK, Ge J, Huo Y. Protocol of the China ST-segment elevation myocardial infarction (STEMI) Care Project (CSCAP): a 10-year project to improve quality of care by building up a regional STEMI care network. BMJ Open. 2019 Jul 17;9(7):e026362. doi: 10.1136/bmjopen-2018-026362. PMID 31320346